CLINICAL TRIAL: NCT05784623
Title: DIGICOG-start: Intérêt et faisabilité de la Technique de DIGItracking Pour Diagnostiquer précocement Les Troubles de la COGnition au Cours de la Vie
Brief Title: Interest and Feasibility of the DIGItracking Technique for the Early Diagnosis of COGnitive Disorders
Acronym: DIGICOG-start
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-162
Record Dates: First submitted 2023-03-01; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Aging
Keywords: digit-tracking; elderly; neurocognitive disorders; usability; user experience
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: User experience — User experience is assessed by validated scales

SUMMARY:
The main objective is to assess the usability of a novel tool of neurocognitive disorders detection, called the Digitracking, by the elderly population. The Digitracking technique is based on the eye tracking concept to assess cognitive decline (Lio et al. 2019). Instead of capturing eye movements, the new device captures the finger trajectory while exploring a blurred picture on a tablet. The usability of such a technology is assessed through objective and subjective metrics, such as the user experience.

DETAILED DESCRIPTION:
Methods for cognitive decline diagnosis in elderly patients using simple, fun and ecological tests remain a major health issue. The objective is the early diagnosis of disorders in order to offer quick management of the decline of cognitive functions.

Eye tracking is a proven technique to study perceptual and cognitive functions in children and adults. It has recently been highlighted that it was also relevant to analyze the perceptual and cognitive functions of elderly people at different stages of neurocognitive disorders. Although very precise, this technique remains restrictive since it requires expensive equipment, technical skills, and long and repetitive tests while the patient stays motionless.

A new approach using the digit-tracking, named Digitrack (Lio et al. 2019), has shown excellent correlation with the eye tracking. The general principle is as follows: a blurred image is displayed on a touchpad screen. This degraded image reproduces the spatial resolution of the peripheral retina. While the patient put his finger on the screen, the area around the finger is unblurred, simulating the foveal region (central region) of the eye. By sliding his finger, the subject moves the unblurred window and can explore the image. The exploration trajectory, like the eye movement trajectory with eye tracking, is recorded and reveals the subjective regions of interest contained in the image which help to assess the user's neurocognitive functions.

The advantage of the Digitrack process is to require a cheap and easy-to-use device to assess the cognitive status of patients in a fun way and close to real conditions.

To date, its usability has not been demonstrated in elderly patients with or without neurocognitive disorders.

The investigators formulate the main hypothesis that patients visiting or hospitalized in the acute care geriatrics department, with or without cognitive disorders, can use the Digitrack process.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 75 years old
* Consultation or hospitalization in geriatrics department
* Subjects who can give written consent to participate in the study

Exclusion Criteria:

* Photosensitive epilepsy
* Uncorrected visual deficiency
* Any significative impairment at the upper limb level preventing from manipulating the device
* Persons deprived of their liberty by administrative or judicial decision, persons under psychiatric care under duress, adults subject to a legal protection measure or unable to express their consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All consecutive patients meeting the eligibility criteria over the study period.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Success rate of the Digitrack use | after 5 minutes of Digitrack use
  The number of patients able to complete the training and evaluation phases with the Digitrack, consisting of the exploration of 3 and at least 20 images respectively.

SECONDARY OUTCOMES:
User experience assessed with the AttrakDiff scale | after 5 minutes of Digitrack use
  The AttrakDiff is composed of 28 items. Each item is presented as a 7-point semantic differential (e.g. "simple - complicated"). The rates range between -3 and 3, 0 being the neutral value. The scores are averaged across the population.
User experience assessed with the modular evaluation of the Components of User Experience (meCUE) questionnaire | after 5 minutes of Digitrack use
  The module II 'emotions' of the meCUE questionnaire is used. It is composed of 8 items. Each item is presented as emotional sentences (e.g. "The product excites me.") and the user rates his agreement with the sentence on a 7-point Likert scale. The scores are averaged across the population
User engagement | after 5 minutes of Digitrack use
  The user engagement is classified according to an internally developped scale including 5 levels : 'interactive', 'constructive', 'active', 'passive', 'disengaged'. The experimenter attributes the level of engagement according to the participant's dominant behavior during the whole experimental procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No
IPD are not planned to be shared with other researchers

REFERENCES:
- [Background] Lio G, Fadda R, Doneddu G, Duhamel JR, Sirigu A. Digit-tracking as a new tactile interface for visual perception analysis. Nat Commun. 2019 Nov 26;10(1):5392. doi: 10.1038/s41467-019-13285-0. PMID 31772154
- [Background] Chi MTH, Wylie R. The ICAP Framework: Linking Cognitive Engagement to Active Learning Outcomes. Educational Psychologist. 2014; 49:219-243.